CLINICAL TRIAL: NCT00457015
Title: EDEMA4: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Assess the Efficacy and Safety of DX-88 (Ecallantide) for the Treatment of Acute Attacks of Hereditary Angioedema
Brief Title: Efficacy Study of DX-88 (Ecallantide) to Treat Acute Attacks of Hereditary Angioedema (HAE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EDEMA4 (DX-88/20)
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Results first posted 2010-05-04 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — ecallantide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DX-88 (ecallantide) (Experimental): DX-88 (ecallantide) 30 mg given as three 10 mg/mL subcutaneous injections.
  Interventions: Drug: ecallantide
- Placebo (Placebo Comparator): Placebo, Phosphate Buffer Saline (PBS), pH 7.0 given as 3 subcutaneous injections.
  Interventions: Drug: Phosphate Buffer Saline (PBS), pH 7.0

INTERVENTIONS:
Drug: ecallantide — dose of 30 mg (10 mg/ml) given as 3 subcutaneous injections.
  Other Names: DX-88
  Arms: DX-88 (ecallantide)
Drug: Phosphate Buffer Saline (PBS), pH 7.0 — given as three 1mL subcutaneous injections.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of DX-88 (ecallantide) versus placebo in the treatment of moderate to severe acute attacks of hereditary angioedema.

DETAILED DESCRIPTION:
This is a randomized placebo-controlled trial.

The study is designed to assess the efficacy and safety of 30 mg subcutaneous ecallantide versus placebo in the treatment of moderate to severe acute attacks of hereditary angioedema. This study is conducted under Special Protocol Assessment with the FDA and is designed to provide pivotal efficacy data on ecallantide. These data are intended to support the marketing authorization of ecallantide in the treatment of acute attacks of hereditary angioedema. Efficacy and safety of ecallantide will be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* 10 years of age or older
* Executed informed consent
* Documented diagnosis of HAE (Type I or II)
* Presentation at the site within 8 hours of patient recognition of an moderate to severe HAE acute attack

Exclusion Criteria:

* Receipt of an investigational drug or device, within 30 days prior to study treatment
* Receipt of non-investigational C1-INH within 7 days of treatment
* Receipt of DX-88 (ecallantide) within 3 days prior to study treatment
* Diagnosis of acquired angioedema (AAE), estrogen-dependent angioedema or drug-induced angioedema (including angiotensin-converting enzyme inhibitor induced angioedema)
* Pregnancy or breastfeeding

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2007-04-01 (Actual); Primary Completion 2008-06-01 (Actual); Study Completion 2008-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (45):
- United States (42):
  - Aaron J. Davis, Scottsdale, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Little Rock Allergy & Asthma Clinic, Little Rock, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Pacific Coast Allergy, Crescent City, California
  - Jacob Offenberger, Granada Hills, California
  - UCLA David Geffen School of Medicine, Department of Medicine, Los Angeles, California
  - Asthma and Allergy Associates, P.C., Colorado Springs, Colorado
  - Christiana Hospital, Newark, Delaware
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami, General Clinical Research Center, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Roberson Allergy and Asthma, West Palm Beach, Florida
  - Family Allergy & Asthma Center, PC, Atlanta, Georgia
  - Allergy Center of Brookstone, Columbus, Georgia
  - University Consultants in Allergy and Immunology, Chicago, Illinois
  - Muncie Allergy Center, Muncie, Indiana
  - Kansas City Allergy & Asthma, Overland Park, Kansas
  - Institute for Asthma and Allergy, Wheaton, Maryland
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - Asthma and Allergy Institute of Michigan, Clinton Township, Michigan
  - Respiratory Medicine Research Institute of Michigan, PLC, Ypsilanti, Michigan
  - Nevada Access to Research and Education Society, Las Vegas, Nevada
  - University of Nevada School of Medicine, Reno, Nevada
  - UMDNJ-New Jersey Medical School, Newark, New Jersey
  - Allergy Partners of Albuquerque, Albuquerque, New Mexico
  - Winthrop University Hospital, Mineola, New York
  - Allergy Partners of Western North Carolina, Asheville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Optimed Research, LLC, Columbus, Ohio
  - Valley Clinical Research Center, Easton, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Asthma Allergy and Pulmonary Associates, Philadelphia, Pennsylvania
  - Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Highlands Allergy and Asthma Center, PC, Bristol, Tennessee
  - The Paull Allergy and Asthma Clinic, P.A., Bryan, Texas
  - AARA Research Center, Dallas, Texas
  - University of Texas Medical School, Galveston, Texas
  - Baylor Clinic, Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Puget Sound Allergy, Asthma, & Immunology, Tacoma, Washington
- Canada (2):
  - Allergy and Asthma Research Center, Ottawa, Ontario
  - University of Toronto, Toronto, Ontario
- Jordan University Hospital, Amman, Jordan

REFERENCES:
- [Derived] Rubinstein E, Stolz LE, Sheffer AL, Stevens C, Bousvaros A. Abdominal attacks and treatment in hereditary angioedema with C1-inhibitor deficiency. BMC Gastroenterol. 2014 Apr 9;14:71. doi: 10.1186/1471-230X-14-71. PMID 24712435
- [Derived] MacGinnitie AJ, Davis-Lorton M, Stolz LE, Tachdjian R. Use of ecallantide in pediatric hereditary angioedema. Pediatrics. 2013 Aug;132(2):e490-7. doi: 10.1542/peds.2013-0646. Epub 2013 Jul 22. PMID 23878046
- [Derived] Sheffer AL, MacGinnitie AJ, Campion M, Stolz LE, Pullman WE. Outcomes after ecallantide treatment of laryngeal hereditary angioedema attacks. Ann Allergy Asthma Immunol. 2013 Mar;110(3):184-188.e2. doi: 10.1016/j.anai.2012.12.007. Epub 2013 Jan 5. PMID 23548529
- [Derived] Li HH, Campion M, Craig TJ, Soteres DF, Riedl M, Lumry WR, MacGinnitie AJ, Shea EP, Bernstein JA. Analysis of hereditary angioedema attacks requiring a second dose of ecallantide. Ann Allergy Asthma Immunol. 2013 Mar;110(3):168-72. doi: 10.1016/j.anai.2012.12.004. Epub 2013 Jan 8. PMID 23548526
- [Derived] Bernstein JA, Shea EP, Koester J, Iarrobino R, Pullman WE. Assessment of rebound and relapse following ecallantide treatment for acute attacks of hereditary angioedema. Allergy. 2012 Sep;67(9):1173-80. doi: 10.1111/j.1398-9995.2012.02864.x. Epub 2012 Jul 5. PMID 22765833
- [Derived] Riedl M, Campion M, Horn PT, Pullman WE. Response time for ecallantide treatment of acute hereditary angioedema attacks. Ann Allergy Asthma Immunol. 2010 Dec;105(6):430-436.e2. doi: 10.1016/j.anai.2010.09.005. Epub 2010 Oct 25. PMID 21130380

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were screened in advance of presenting with an HAE attack but were randomized only upon attack.
Groups:
- KALBITOR (Ecallantide): KALBITOR (ecallantide, DX-88) 30 mg given as three 10 mg/mL subcutaneous injections.
Period: Overall Study
Arm/Group | KALBITOR (Ecallantide) | Placebo
Started | 48 | 48
Completed | 48 | 47
Not Completed | 0 | 1
Not completed — Left study site against medical advice | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KALBITOR (Ecallantide) | Placebo | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (13.12) | 38.0 (12.19) | 37.5 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 28 | 65
  Male | 11 | 20 | 31
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47 | 48 | 95
  Canada | 1 | 0 | 1
Symptom Complexes at Baseline [Number; unit: symptom complexes] — More than one baseline symptom complex could be reported per patient; hence the number of complexes is greater than the number of patients in each group. Patient were to have at least one symptom complex that was moderate or severe. The total number of symptom complexes was 155.
  symptom complexes
    Internal Head/Neck | 8 | 13 | 21
    Stomach/GI | 18 | 27 | 45
    Genital/Buttocks | 6 | 5 | 11
    External Head/Neck | 14 | 9 | 23
    Cutaneous | 34 | 21 | 55

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Symptom Complex Severity (MSCS) Score at 4 Hours Post-dose
Description: The Mean Symptom Complex Severity (MSCS) score is a validated, comprehensive point-in-time measure of symptom severity. At baseline and 4 hours, patients rated the severity on a categorical scale (0 = normal, 1 = mild, 2 = moderate, 3 = severe) for symptoms at each affected anatomical location. Ratings were averaged to obtain the MSCS score. A decrease in MSCS score reflected an improvement in symptoms; clinically meaningful improvement was indicated by a reduction in the score of 0.30 or more.
Time Frame: baseline, 4 hours post-dose
Population: Patients were excluded from the analysis if they did not have data for the endpoint being analyzed. Reasons for patients being excluded are for ecallantide: 1 patient treated for severe upper airway compromise; for placebo: 3 patient treated for severe upper airway compromise and 3 patients with missing 4-hour data. Best score=0.0; worst score=3.0.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | KALBITOR (Ecallantide) | Placebo
Number analyzed (Participants) | 47 | 42
units on a scale
  MSCS Score at baseline | 2.2 (0.50) | 2.0 (0.35)
  MSCS Score at 4 hours post-dose | 1.4 (0.75) | 1.6 (0.77)
  Change from baseline in MSCS at 4 hours post-dose | -0.8 (0.63) | -0.4 (0.82)
Statistical Analysis 1: Comparison: KALBITOR (Ecallantide) vs Placebo; The primary efficacy analysis compared the change from baseline in MSCS Score at 4 hours post-dosing for patients treated with ecallantide and placebo. Treatment effect was assessed by the nonparametric Blocked Wilcoxon Rank Sum test because of an assumed non-normal distribution; Test type: Superiority or Other; p = 0.010, Blocked Wilcoxon rank sum test — No adjustment was made for multiple comparisons. Treatment effect will be deemed statistically significant if the coefficient for the treatment group within the statistical model is significant at level 0.05

2. Secondary Outcome: Treatment Outcome Score at 4 Hours Post-Dose
Description: Treatment Outcome Score (TOS) is a validated, comprehensive measure of symptom response to treatment. At 4 hours , patient assessment of response characterized by their change from baseline in symptom severity and collected by anatomic site of attack involvement, was recorded on a categorical scale (significant improvement [100; best value]to significant worsening [-100; worst value]). Clinically meaningful improvement was indicated by a TOS of 30 or higher.
Time Frame: 4 hours post-dose
Population: Patients were excluded from this analysis if they did not have data for the endpoint being analyzed. The reasons for patients being excluded from this analysis are for ecallantide: 1 patient treated for severe upper airway compromise and for placebo: 3 patient treated for severe upper airway compromise and 3 patients with missing 4-hour data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | KALBITOR (Ecallantide) | Placebo
Number analyzed (Participants) | 47 | 42
units on a scale | 53.4 (49.70) | 8.1 (63.18)
Statistical Analysis 1: Comparison: KALBITOR (Ecallantide) vs Placebo; The analysis compared the TOS at 4 hours post-dosing for patients treated with ecallantide and placebo. Treatment effect was assessed by the nonparametric Blocked Wilcoxon Rank Sum test because of an assumed non-normal distribution; Test type: Superiority or Other; p = 0.003, Blocked Wilcoxon rank sum test — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Patients With Significant Improvement in Overall Response
Description: Patients were to be asked to perform an overall response assessment at intervals during the first 4 hours post-dose. Assessments were to be made relative to baseline (ie, immediately before initial dosing) using a 5-category scale. Categories were: significant improvement = "a lot better or resolved"; improvement = "a little better"; same = response unchanged; worsening = "a little worse"; significant worsening = "a lot worse". Significant improvement is the first time that a patient responded to the overall response assessment as "a lot better or resolved."
Time Frame: 4 hours post-dose
Population: The time to significant improvement is not provided in this display as the estimated median times were not reached by 240 minutes. Instead, the number of patients with significant improvement is provided per treatment arm.
Measure: Number; unit: participants
Arm/Group | KALBITOR (Ecallantide) | Placebo
Number analyzed (Participants) | 48 | 48
participants | 22 | 12
Statistical Analysis 1: Comparison: KALBITOR (Ecallantide) vs Placebo; Kaplan-Meier analysis using the Log-Rank test was used to compare the time distribution between the 2 treatment groups; Test type: Superiority or Other; p = 0.102, Log Rank — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Patients With a Successful Response at 4 Hours Post-dosing, Based on the Change From Baseline in the MSCS Score
Description: A successful response was defined as improvement in existing laryngeal symptom complex,stabilization of an existing peripheral symptom complex, or a change from baseline in the MSCS score at 4 hours of at least -1.0.
Time Frame: baseline, 4 hours post-dosing
Population: Diary information was not available for 1 patient in the placebo arm. This patient was considered not evaluable and excluded from the analysis.
Measure: Number; unit: participants
Arm/Group | KALBITOR (Ecallantide) | Placebo
Number analyzed (Participants) | 48 | 47
participants | 45 | 28

5. Secondary Outcome: Proportion of Patients Maintaining a Significant Improvement in Overall Response Through 24 Hours
Description: Maintenance of significant improvement was defined as achieving and maintaining a significant improvement in overall response through 24 hours after dosing. Patient response categories were: significant improvement = "a lot better or resolved"; improvement = "a little better"; same = response unchanged; worsening = "a little worse"; significant worsening = "a lot worse".
Time Frame: 24 hours post-dosing
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | KALBITOR (Ecallantide) | Placebo
Number analyzed (Participants) | 48 | 47
participants | 21 | 10

ADVERSE EVENTS:
Time Frame: up to 7 days post-dose
Description: For patients that were given an open-label dose of ecallantide for severe upper airway compromise or failed or incomplete response, or relapse, all adverse events occurring prior to open-label dosing are included in the following tables where all patients are presented in the double-blind, randomized treatment groups.
Arm/Group | KALBITOR (Ecallantide) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/48 | 3/48
Other Adverse Events (participants affected / at risk) | 5/48 | 9/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KALBITOR (Ecallantide) (N=48) | Placebo (N=48)
Hereditary angioedema (Congenital, familial and genetic disorders) | 0 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | KALBITOR (Ecallantide) (N=48) | Placebo (N=48)
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Headache (Nervous system disorders) | 2 | 5
Nausea (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Dyax agreements vary, but Dyax will not prohibit any investigator from publishing. Dyax reviews publications prior to public release and can request deferral by up to 60 days beyond the proposed publication date if necessary to preserve its intellectual property. Dyax can request changes to publications to remove non-study-related confidential information. Dyax can also request deferral of single-center publications until after disclosure of the clinical trial's primary publication.